CLINICAL TRIAL: NCT05103774
Title: Thyroid Functions in Children With Congenital Heart Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hend Abdelrahim Saber, Resident doctor at Pediatric department Sohag University hospital, Sohag University
Other Study IDs: Soh Med-21-10-24
Record Dates: First submitted 2021-10-18; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Value of Thyroid Functions in Children With Congenital Heart Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: children exposed to any type of radiation or contrast: Group A: children exposed to any type of radiation or contrast
  Interventions: Diagnostic Test: T3-T4-TSH
- Group B : children not exposed to an type of radiation or contrast: Group B : children not exposed to an type of radiation or contrast
  Interventions: Diagnostic Test: T3-T4-TSH

INTERVENTIONS:
Diagnostic Test: T3-T4-TSH — thyroid function tests

SUMMARY:
Thyroid hormone is critical for normal neurocognitive development in young infants, and even transient hypothyroidism can cause adverse neurodevelopmental outcomes. In a population of infants with CHD who already bear a high risk of long-term developmental delay, detection of hypothyroidism, even of a transient nature, may be even more consequential, and routine periodic monitoring of thyroid function may be necessary to reduce the risk of neurodevelopmental disabilities

ELIGIBILITY:
Inclusion Criteria:

* All children since birth up to age of 12 years old including both genders diagnosed to have CHD exposed to radiation, contrast or not.

Exclusion Criteria:

* above 12 years old

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Place of the study: Sohag University Hospital (pediatrics department -cardiology unit).
  * Sample size the whole sample size will be at least 100 child diagnosed as CHD divided equally into two groups (group A and B) Group A: children exposed to any type of radiation or contrast Group B : children not exposed to an type of radiation or contrast
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of thyroid function in children with congenital heart diseases at Sohag University hospital | One year
  Thyroid function tests will be obtained from children with congenital heart diseases as will as the control group

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided